CLINICAL TRIAL: NCT01973530
Title: Comparison of the Analgesic Efficacy of Continuous Femoral Nerve Block and Adductor Canal Block With Steroid Adjuvant in Patients Undergoing Total Knee Arthroplasty
Brief Title: Comparison of Femoral Nerve Catheter and Adductor Canal Block With Steroid Adjuvant in Total Knee Replacement (TKR)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Hui Kit Man Grace, Associate Consultant, Dept of Anaesthesia and Operating Services, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHJRC_HK_TKR_Study_2014
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis
Keywords: femoral nerve block; adductor canal block; steroid; total knee replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adductor canal block (Active Comparator): Continuous adductor canal block and single shot posterior tibial nerve block under ultrasound guidance and using nerve stimulating needle (bolus: 0.5% Ropivacaine 10-15ml with dexamethasone 4mg ;with single shot posterior tibial nerve block (8-10ml 0.5% ropivacaine)
  Interventions: Procedure: adductor canal block
- continuous femoral nerve block (Other): Femoral nerve catheter inserted under ultrasound guidance using nerve stimulating needle administering ropivacaine bolus 10-15ml and infusing 0.2% ropivacaine at 4-6ml/h; plus a single shot posterior tibial nerve block under ultrasound guidance and use of nerve stimulating needle
  Interventions: Procedure: femoral nerve block

INTERVENTIONS:
Procedure: adductor canal block — Continuous adductor canal block and single shot posterior tibial nerve block under ultrasound guidance and using nerve stimulating needle (bolus: 0.5% Ropivacaine 10-15ml with dexamethasone 4mg ;with single shot posterior tibial nerve block (8-10ml 0.5% ropivacaine)
  Arms: adductor canal block
Procedure: femoral nerve block — Femoral nerve catheter inserted under ultrasound guidance using nerve stimulating needle administering ropivacaine bolus 10-15ml and infusing 0.2% ropivacaine at 4-6ml/h; plus a single shot posterior tibial nerve block under ultrasound guidance and use of nerve stimulating needle
  Arms: continuous femoral nerve block

SUMMARY:
We hypothesize continuous adductor canal block with steroid adjuvant would offer no inferior analgesics and rehabilitation ability than continuous femoral nerve block for postoperative patients receiving total knee arthroplasty.

DETAILED DESCRIPTION:
A total of 80 patients who will undergo total knee arthroplasty will be randomized into two groups:

Treatment groups Treatment details Femoral Group (40 patients) Continuous femoral nerve block (bolus: 0.5% Ropivacaine 10-15 ml ; infusion of 0.15 % Ropivacaine 4-6ml/h) Adductor Group (40 patients) Adductor canal block with steroid adjuvant (bolus: 0.5% Ropivacaine 10-15ml; Dexamethasone 4mg) (Total 80 patients will be recruited)

* All patients will receive single shot tibial nerve block with local anaesthetics (0.5% Ropivacaine 5-8ml) before surgery for analgesia of posterior knee.
* All patients will receive the same preemptive and postoperative multimodal medications for perioperative analgesia.
* All groups will receive standardized method of spinal anaesthesia and standardized method of intraoperative sedation for the surgery.
* Intravenous patient controlled analgesia (PCA) with morphine will be given for 48h to patient as rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis
* Scheduled for elective total knee arthroplasty
* Signed written informed consent
* Planned use of spinal anaesthesia
* Cognitive sound to use assessment tools

Exclusion Criteria:

* Patients refusing to give consents
* Scheduled for revision total knee replacement
* Patient outside range of 30 to 80 yrs old
* Non-chinese population
* Cognitive impairment/ inability to use the outcome assessment tools
* Contraindications to regional anesthesia
* severe cardiovascular disease (unstable angina, second or third degree heart block)
* pre-existing neurologic disease including psychiatric disorder
* drug abuser
* Pre-operative history of neurological abnormality in the ipsilateral leg e.g. history of stroke, neurogenic pain or previous nerve injury.
* Allergy or contraindication to drugs used in this study: morphine, Non-steroidal anti-inflammatory drugs (NSAID) such as ketorolac , diclofenac, dihydrocodeine, local anaesthetics (lignocaine, ropivacaine, bupivacaine), epinephrine
* Moderate or severe renal impairment (serum creatinine > 160 micromol/l)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
PCA morphine or pain rescuer consumption at 24h and 48h postoperative | 24h and 48h postoperative
Postoperative pain score (visual analogue scale 0-10) at 6h,12h, 24h,48h, 72h after surgery | 6h,12h, 24h,48h, 72h after surgery
Quadriceps strength at 24h, 48h, 72h postoperative | 24h, 48h, 72h postoperative
  using dynamometer (measure in Newton/centimeter square)

SECONDARY OUTCOMES:
Patient satisfaction score (0-4) | upon discharge
Incidence of side effects and complications at postoperative day 0- 4 postoperative | postoperative period 0-96 hr postoperative
Length of Stay in hospital 6. Length of Stay in hospital length of hospital stay | upon discharge
postoperative nausea or vomiting | 0-72h
postoperative pruritis | 0-72h
Haemastix on call and every 8 hours after surgery for postoperative 24hours for patients | on call and every 8 hours after surgery for postoperative 24h

CONTACTS AND LOCATIONS:
Overall Officials: Eric So, FHKCA FHKAM, Principal Investigator — Queen Elizabeth Hospital, Hospital Authority
Locations (1):
- Joint Replacement Center, Buddhist Hospital, Kowloon, Hong Kong